CLINICAL TRIAL: NCT02971033
Title: Ezetimibe as a Safe and Efficacious Treatment for Chronic Hepatitis C
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Funding ended
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INFA-015-16S
Record Dates: First submitted 2016-10-21; First posted 2016-11-22 (Estimated); Results first posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Chronic Hepatitis C
Keywords: hepatitis C virus; antiviral treatment; viral entry inhibitor; mathematical modeling
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- 20mg/day ezetimibe (Experimental): 20mg/day ezetimibe
  Interventions: Drug: 20mg ezetimibe
- 40mg/day ezetimibe (Experimental): 40mg/day ezetimibe
  Interventions: Drug: 40mg ezetimibe

INTERVENTIONS:
Drug: 20mg ezetimibe — Participants assigned to this intervention will receive 20mg per day of ezetimibe for 12 weeks.
  Other Names: 20mg Zetia
  Arms: 20mg/day ezetimibe
Drug: Placebo — Participants assigned to this intervention will receive placebo every day for 12 weeks
  Arms: placebo
Drug: 40mg ezetimibe — Participants assigned to this intervention will receive 40mg per day of ezetimibe for 12 weeks.
  Other Names: 40mg Zetia
  Arms: 40mg/day ezetimibe

SUMMARY:
To address the need for more affordable hepatitis C virus (HCV) antivirals with high barriers to viral resistance and strategies to shorten the current treatment duration, the goal is to develop affordable therapeutic regimens to prevent HCV entry/spread and test the efficacy of those inhibitors for treating HCV infection. The investigators recently discovered that a major cholesterol uptake receptor is required for HCV entry into hepatocytes and that there is already an FDA-approved drug that inhibits cholesterol uptake by this receptor. Importantly the same drug also potently blocks HCV entry in human liver cells both in cell culture and in a small animal model. Further, looking back at people who were previously treated for HCV infection, the investigators found treatment response to be better (i.e. larger viral log reduction) in patients who happened to be taking ezetimibe (EZE). Hence, the objective of this study is to assess whether the FDA-approved drug (ezetimibe) is useful for the treatment of chronic HCV. The investigators predict that when administered as monotherapy ezetimibe will reduce HCV viremia perhaps allowing for viral clearance and that when included in combination treatment regimens that EZE will increase HCV decline resulting in faster viral clearance (i.e. shorter/cheaper direct-acting antiviral [DAA] therapy). To test these hypotheses, the investigators will execute the following aims: (1) Assess the efficacy of EZE monotherapy in chronically HCV infected and predict time to cure; (2) Assess the efficacy of EZE as an adjunct therapy in chronically HCV infected patients undergoing currently approved HCV DAA treatment.

DETAILED DESCRIPTION:
To address the need for more affordable HCV antivirals with high barriers to viral resistance and/or strategies to shorten the current treatment duration, the goal is to develop affordable therapeutic regimens to prevent HCV entry/spread and test the efficacy of those inhibitors for treating HCV infection. The investigators recently discovered that the Niemann-Pick C1 Like-1 (NPC1L1) cellular cholesterol uptake receptor is required for HCV entry into hepatocytes and that ezetimibe, an FDA-approved drug that inhibits NPC1L1-mediated cholesterol uptake potently blocks HCV entry in human hepatoma cells and human hepatocytes transplanted into urokinase-type plasminogen activator-severe combined immunodeficiency (uPA-SCID) mice. Further, retrospective analysis of the National VA database using multivariable logistic regression models to control for age, sex, race, alcohol use, drug use, and other co-morbidities, the investigators found HCV prevalence to be lower (p <.001) and interferon/ribavirin (IFN/RBV) treatment response to be better (i.e. larger viral log reduction) in patients taking ezetimibe. Hence, the specific objective of this application is to assess the efficacy of EZE for the treatment of chronic HCV. Based on preliminary in vitro, in vivo, clinical retrospective data and HCV/DAA modeling, the investigators hypothesize that when administered as monotherapy EZE will reduce HCV viremia perhaps allowing for viral clearance and that when included in combination treatment regimens that EZE will augment 2nd phase HCV decline resulting in faster viral clearance (i.e. shorter/cheaper DAA therapy). To test these hypotheses, the investigators will execute the following aims: (1) Assess the efficacy of EZE monotherapy in chronically HCV infected and predict time to cure; (2) Assess the efficacy of EZE as an adjunct therapy in chronically HCV infected patients undergoing currently approved HCV DAA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males/females 18 - 70 yrs of age
* Serum HCV RNA >2,000 IU/ml
* Hepatitis C genotype 1
* Other causes of chronic liver disease excluded by appropriate clinical, laboratory, or histologic evaluation
* The following hematological criteria must be met:

  * Hemoglobin > 12 g/dl
  * Absolute neutrophil count (ANC) > 1.0x109 /L
  * Platelets 150 x 108 /L (i.e normal)
* Serum creatinine <1.5 times the upper limit of normal (ULN) at screening.
* Fasting blood sugar normal for non-diabetics or hemoglobin A1C < 8.5% with diabetes
* Women of childbearing potential must have a negative pregnancy test prior to receiving treatment. Sexually active women must take adequate precautions to prevent pregnancy during the study. Pregnancy tests will be done at the final clinic visits and every 4 weeks
* Patient provides written informed consent

Exclusion Criteria:

* Evidence of liver disease other than HCV:

  * Antinuclear antibodies (ANA) >1:160
  * Active alcoholic liver disease.
  * Hepatitis B surface antigen positive
  * Hemochromatosis
  * Wilson disease
  * Alpha-1-antitrypsin deficiency
  * Recent hepatotoxic drug exposure
  * Cirrhosis with complications of portal hypertension including esophageal varices (> grade 1 by endoscopy), ascites, or hepatic encephalopathy, or bilirubin >2.0 mg/dl
* Patients with advanced fibrosis (defined herein as decompensated cirrhosis, FIB4 > 2.5, platelet count <150 x 103/uL, clinical or radiographic evidence of cirrhosis)
* Extrahepatic manifestations of liver disease or HIV co-infection
* Use of fibric acid, Fenofibrate or cholestyramine
* Active substance abuse including, but not limited to alcohol or i.v./inhaled drugs
* Use of chemotherapy or systemic steroid therapy within 30 days prior to enrollment
* Pregnancy, females who are breast feeding, or females of child bearing potential who are not using adequate birth control measures
* History of a medical condition that could interfere with participation or completion of the protocol
* Organ transplant recipient
* History of hypersensitivity to ezetimibe

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L. Uprichard, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients are enrolled, but then are not randomized until they pick up clinical and study medication with the investigational pharmacist at a subsequent visit. As such, one can be enrolled but never randomized if they patient does not return for the medication.
Groups:
- Placebo: placebo
  Placebo: Participants assigned to this intervention will receive placebo every day for 8 weeks
- 20mg/Day Ezetimibe: 20mg/day ezetimibe
  20mg ezetimibe: Participants assigned to this intervention will receive 20mg per day of ezetimibe for 8 weeks.
- 40mg/Day Ezetimibe: 40mg/day ezetimibe
  40mg ezetimibe: Participants assigned to this intervention will receive 40mg per day of ezetimibe for 8 weeks.
Period: Overall Study
Arm/Group | Placebo | 20mg/Day Ezetimibe | 40mg/Day Ezetimibe
Started | 1 | 1 | 0
Completed | 1 | 1 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: no patients were randomized to 40mg/day ezetimibe group
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 20mg/Day Ezetimibe | 40mg/Day Ezetimibe | Total
Number analyzed (Participants) | 1 | 1 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 0 | 2
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  non-hispanic White | 0 | 1 | 0 | 1
  non-hispanic Black | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 1 | 0 | 2
HCV RNA [Mean (Full Range); unit: International Units per mL] — HCV RNA is measured by clinical laboratories by reverse transcription quantitative PCR, which measures the number HCV genomes present. The results are reported as international units per milliliter (IU/mL). Higher HCV IU means higher levels of HCV in the blood.
  International Units per mL | 4030000 [4030000 to 4030000] | 5860000 [5860000 to 5860000] |  | 4945000 [4030000 to 5860000]
alanine transaminase (ALT) [Mean (Full Range); unit: Units/Liter] — Participants will have their ALT levels measured in units per liter (U/L) at baseline. ALT ranges from 0 to infinity with higher levels of ALT indicating liver cells damage.
  Units/Liter | 109 [109 to 109] | 105 [105 to 105] |  | 107 [107 to 109]

OUTCOME MEASURES:

1. Primary Outcome: Change in Viral Load
Description: Participants will have their HCV-RNA measured in international unit per milliliter at baseline and 8 weeks. HCV RNA international unit per milliliter ranges from 0 to infinity, with higher levels indicating HCV positivity. The change in international unit per milliliter will be compared among the three intervention groups (i.e., placebo or control cohort, those assigned to 20mg ezetimibe per day, and 40mg ezetimibe per day). Change is calculated based on 8 weeks minus baseline (0 weeks).
Time Frame: 0 weeks, 8 weeks
Population: Participants who were enrolled, were not randomized until they received their study medication. No one was randomized to the 40mg/day arm
Measure: Mean (Full Range); unit: international units per milliliter
Arm/Group | Placebo | 20mg/Day Ezetimibe | 40mg/Day Ezetimibe
Number analyzed (Participants) | 1 | 1 | 0
international units per milliliter | -4030000 [-4030000 to -4030000] | -5860000 [-5860000 to -5860000] |

2. Primary Outcome: Second Phase Slope
Description: HCV declines in a biphasic manner under HCV treatment. Here we are measuring the slope (i.e., rate) at which HCV is declining during the second slower phase of viral decline.
Time Frame: 3 days through 4 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: log(copies/mL)/day
Arm/Group | Placebo | 20mg/Day Ezetimibe | 40mg/Day Ezetimibe
Number analyzed (Participants) | 1 | 1 | 0
log(copies/mL)/day | .90 [.90 to .90] | .98 [.98 to .98] |

3. Secondary Outcome: Change in Alanine Aminotransferase (ALT)
Description: Participants will have their ALT levels measured in units per liter (U/L) at baseline and 8 weeks. ALT ranges from 0 to infinity with higher levels of ALT indicating hepatocyte death. The change in ALT levels will be compared among the three intervention groups (i.e., placebo or control cohort, those assigned to 20mg ezetimibe per day, and 40mg ezetimibe per day).
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: units per Liter
Arm/Group | Placebo | 20mg/Day Ezetimibe | 40mg/Day Ezetimibe
Number analyzed (Participants) | 1 | 1 | 0
units per Liter | -75 [-75 to -75] | -73 [-73 to -73] |

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: there were no patients randomized to the 40mg/day ezetimibe arm
Arm/Group | Placebo | 20mg/Day Ezetimibe | 40mg/Day Ezetimibe
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
1. A major limitation is that the study was that it was interrupted by the CoVID-19 pandemic and then was terminated early leading to small numbers of subjects analyzed. It is not possible to derive conclusions comparing the single patients enrolled in arms 1 and 2.
2. The patient in arm 2 had study medication remaining at the first pill count indicating that EZE dosing was lower than 20mg/day during at least part of the treatment period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT02971033/Prot_SAP_000.pdf